CLINICAL TRIAL: NCT04027582
Title: Role of Simulators to Assess Simulator-Based Entrusted Professional Activity in Fiber-optic Intubation and Transfer-ability to Clinical Assessment of Anesthesia Trainees in the Competency By Design Residency Program
Brief Title: Comparing Simulators Used in Fiber-optic Intubation Training Among Anesthesia Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Eric You-Ten, Associate Professor Anesthesia, Mount Sinai Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 19-0020-A
Record Dates: First submitted 2019-07-18; First posted 2019-07-22 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Fiber-optic Intubation
Keywords: ORSIM; Entrustable Professional Activity

STUDY DESIGN:
Intervention Model Description: This is a 2-arm comparison study to be conducted at Mount Sinai Hospital, Toronto.
  After written informed consent, participants will be randomized to the low fidelity simulator (LFS n=15) and the high- fidelity simulator (ORSIM, n=15). Participants consist of anesthesia 1st - 2nd year residents in the Competency-based Medical Education Anesthesia Residency program, Emergency Medicine Residents, Family Practice Anesthetists and Emergency Residents with less than five prior experiences in fiberoptic intubations.
Who Masked: Outcomes Assessor
Masking Description: The assessors of the video-recorded Simulator EPA and Patient EPA will be blinded as to what group the resident was allocated to . i.e the Low fidelity simulator group or the high fidelity simulator group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Fidelity Simulator - Wooden block (Active Comparator): This simulator consists of a simple series of wooden panels with holes. The resident learns how to manipulate the fiberoptic bronchoscope through the holes.
  Interventions: Other: didactic teaching and simulator practice
- High fidelity Simulator - ORSIM (Active Comparator): The ORSIM® bronchoscopy is a virtual reality simulator (Airway Simulation Limited, Auckland, New Zealand). It consists of hardware and software components that interact to create a high-fidelity virtual reality simulation. A replica fiberoptic scope is advanced by the resident through a desktop sensor, which is connected to a laptop computer. The laptop software program provides a virtual airway in which the user must navigate the probe.
  Interventions: Other: didactic teaching and simulator practice

INTERVENTIONS:
Other: didactic teaching and simulator practice — the trainee will undergo didactic teaching on fiber-optic intubation followed by hands on practice on their assigned simulator

SUMMARY:
Thirty residents in Anesthesia, year one and year two ,and Emergency Medicine Residents, and Family Practice Anesthetists and Emergency residents will undergo teaching in fiber-optic intubation. One half of the group will be randomized to a low fidelity simulator which consists of a wooden block with a series of holes, and the other to a high fidelity simulator, called the ORSIM , which provides a computerised model of the airway. They will practice the procedural skill of fiber-optic intubation on their assigned simulators. Cumulative sum method (CUSUM) learning curves and procedural Entrusted Professional Activities will be obtained for each resident on their assigned simulator. Following this , all residents will undergo a procedural entrusted professional activity with regard to fiber-optic intubation on a low risk , consented patient. The results of the learning curves, Simulator entrusted professional activity and Patient entrusted professional activity will be compared to assess if there is a difference between the low fidelity and high fidelity simulator groups.

DETAILED DESCRIPTION:
Fiber-optic intubation(FOI) involves using a thin flexible scope to navigate a breathing tube into a patient's trachea. It is an important skill, as it is required in situations where the breathing tube cannot be inserted using traditional methods. It is a lifesaving skill in terms of securing the 'the difficult airway', in emergency and elective situations. The National Audit Project 4 (NAP4, the largest study on major airway complications in the operating room, emergency department and intensive care unit) have identified the omission of FOI when indicated as a major contributor to airway morbidity and mortality . Recommendations from NAP4 included ensuring anesthesiologists are trained in the use of FOI.

Medical training in Canada and globally is undergoing a major transformation to competency-based medical education (CBME). Within the next decade, all residency programs in Canada will be following a competency-based curriculum, as mandated by the Royal College of Physicians and Surgeons of Canada (Royal College) and the College of Family Physicians of Canada. CBME emphasizes the demonstration of competence in skills and abilities deemed essential for future practice and de-emphasizes time and duration .

While competence is assessed by several metrics in CBME, the entrustable professional activities (EPAs)framework is one approach to assessment. EPAs are specific tasks in the clinical environment that a supervisor will delegate to a resident once sufficient competence has been demonstrated .

Competency-based medical education(CBME) requires residents to demonstrate competency in key skills; simulators have an important role in facilitating this learning in a safe environment without harming patients. Currently, little is known on the role of simulators on acquiring competence of Fiber-optic intubation and assessment of simulator-based Entrusted Professional Activity (EPA) and transfer-ability to patient -based EPA.

The focus of the study is the learning aspect with regards to fiber-optic intubation.

The hypothesis is that simulator-based EPA is transferable to clinical-based EPA and that clinical performance is better after training with a high -fidelity simulator.

Methods:

This is a 2-arm comparison study to be conducted at Mount Sinai Hospital, Toronto.

After written informed consent, resident participants will be randomized to the low fidelity simulator (LFS n=15) and the high- fidelity simulator (ORSIM, n=15). Participants consist of anesthesia 1st - 2nd year residents in the Competency-based Medical Education Anesthesia Residency program, Emergency Medicine Residents, Family Practice Anesthetists and Emergency Medicine Residents, with less than five prior experiences in fiberoptic intubations.

The resident will undergo a teaching intervention consisting of a didactic Power-point presentation and video on FOI, {https://www.youtube.com/watch?v=wDLrRHS7Urw}, followed with hands-on practice on the LFS or ORSIM. The didactic teaching will be group based, but the hands-on simulator practice will be one to one.

Generating Learning Curve (CUSUM) for Competence:

After the teaching session, the resident participant will generate a learning curve for a series of fiberoptic intubations on the respective simulator using the cumulative sum method (CUSUM).The resident will be allowed 20 attempts. Residents will be considered simulator-competent if they reach 90% success rate.

Simulator-based Entrusted Professional Activity (EPA) Assessment:

Within one week later the resident will be assessed to complete an EPA on fiber-optic intubation using their assigned simulator. Each performance will be video-recorded for data analysis by the research assistant.

Transfer to Clinical-based EPA Assessment:

Thereafter and within two weeks, the resident will then perform a fiber-optic intubation on an anesthetized patient in the Operating Room. The fiberoptic intubation on a patient will be limited to a maximum of 8 minutes since this is the apnea time where desaturation (hypoxia) will occur in a patient induced with general anesthesia and muscle paralysis who underwent adequate pre-oxygenation. .

Written informed consent will be obtained from each patient.

The performance of the Simulator based EPA and clinical EPA will be video-recorded. No patient or resident identifiers will be recorded, the patient's eyes will be covered with a surgical green towel, leaving the mouth and nose exposed to bag mas ventilate, the camera will focus on the resident's hands.

Two experienced observers will grade the intubations using a validated checklist and global rating scale. They will be blinded to the group allocation.

An experienced anesthetist not involved in the study will be present in the operating room to assist the resident and take over the intubation if they deem necessary for patient safety.

The total time commitment for the resident will be a maximum of 2 hours.

ELIGIBILITY:
Inclusion Criteria:

Participants:

* Anesthesia first and second year residents in the Competency-based Medical Education Anesthesia Residency program
* They must have less than five prior experiences in fiber-optic intubation.

Patient inclusion criteria:

* American Society of Anaesthesiologists classification one and two
* Normal airway anatomy.

Exclusion Criteria:

Patient exclusion criteria:

* Emergency surgery
* Risk of aspiration
* History of Malignant Hyperthermia
* History of succinylcholine Apnea.
* American Society of Anaesthesiologists grade greater than two
* Abnormal airway anatomy
* Morbid obesity
* Difficult bag mask ventilation.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Cumulative sum learning curve | eight minutes
  Primary outcome: Cumulative sum learning curves will be generated as the primary outcome measure as the number of fiber-optics done on each respective simulator to achieve competence, defined as 90% success rate in a series of fiber-optic intubations. Each successful attempt on the respective simulator must be completed within eight minutes (ie apnea time)

SECONDARY OUTCOMES:
Time | eight minutes
  Fiber-optic scope entry to mouth to successful pass through vocal cords, 1-2 cm above the carina.

OTHER OUTCOMES:
Simulator Entrusted Professional Activity score | Eight minutes
  One for entrusted and Zero for non-entrusted
Patient Entrusted Professional Activity score | Eight Minutes
  One for entrusted and Zero for non-entrusted
Checklist score on fiber-optic intubation on patient | Eight Minutes
  validated checklist on fiber-optic intubation Checklist for Intraoperative Fiberoptic Orotracheal Intubation Performance If Done Correctly select yes or no
  1. Holds control section correctly in one hand with thumb positioned for flexion and extension control, and index finger for suction
  2. Focuses scope using appropriate external object
  3. Controls tip of scope with other hand
  4. Introduces bronchoscope into mouth centered
  5. Maneuvers bronchoscope through oropharynx and visualizes cords
  6. Passes cords
  7. Continues insertion of bronchoscope to level of carina
  8. Passes endotracheal tube a-traumatically
  9. Reconfirms vision of carina after endotracheal tube in situ 10 Removes bronchoscope smoothly endo-tracheal tube
Global Rating Score on fiber-optic intubation on patient | Eight Minutes
  Global Rating Scale of Intraoperative Fiber-optic Orotracheal Intubation Performance The scale is from One to Five. One is the lowest score and five is the highest score.
  1. Respect for tissue.
  2. Time and motion .
  3. Knowledge of Instruments.
  4. Flow of Procedure.
  5. Use of Assistants.
  6. Knowledge of procedure.
  7. Overall Performance.

CONTACTS AND LOCATIONS:
Overall Officials: Kong Eric You-Ten, MD PhD FRCPC, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication